CLINICAL TRIAL: NCT07127510
Title: Measurement of Brain NAD Levels in Alzheimer's Patients and Control Subjects by 1H-MRS
Brief Title: Brain NAD in Alzheimer's Disease
Acronym: ALZNAD
Status: Recruiting | Type: Observational
Sponsor: Florida Atlantic University (Other)
Responsible Party: Principal Investigator, Corinne Lasmezas, Professor, Florida Atlantic University
Other Study IDs: IRB2504137
Record Dates: First submitted 2025-08-11; First posted 2025-08-17 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Alzheimer Disease (AD)
Keywords: NAD; Alzheimer Disease (AD)
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Whole blood, plasma and urine
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Alzheimer's disease group: People diagnosed with Alzheimer's disease
- Control group: People without Alzheimer's disease

SUMMARY:
The goal of this observational study is to learn about the levels of nicotinamide adenine dinucleotide (NAD) in the brains of people with Alzheimer's disease. The study aims to determine if brain NAD levels are lower in people with Alzheimer's disease compared with people of the same age group who do not have Alzheimer's disease.

Participants with or without Alzheimer's disease will have a brain imaging session where NAD will be measured using magnetic resonance spectroscopy (MRS). Eight months later, they will have a second, similar, brain imaging session.

ELIGIBILITY:
Inclusion Criteria:

* Participants are able to come to the Florida Atlantic University Clinical Research Unit, are verbal and ambulatory.
* Age 65 to 80 included.
* People with Alzheimer's disease (AD): AD diagnosis established by the person's physician according to the following criteria: clinical diagnosis AND either positive amyloid PET-scan or FDA-approved positive CSF or blood test.

Exclusion Criteria:

* Under the age of 65 or over the age of 80.
* Advanced dementia such that the person would require sedation for undergoing an MRI scan.
* Receiving anti-amyloid intravenous treatments Leqembi or Kinsula.
* Having an MRI-incompatible pacemaker or other MRI-incompatible hardware (e.g. comprising a metallic part).
* Having a history of seizures.
* Working at night.
* Having cancer or having been diagnosed with cancer within the last 5 years (excluding superficial squameous or basal cell cancer).
* People with no AD: MoCA test result lower than 26.

Ages: 65 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: Primary care clinic, community.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2025-12-15 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Brain NAD | At enrollment and 8 months after enrollment
  NAD levels measured by 1H-MRS

CONTACTS AND LOCATIONS:
Overall Officials: Corinne Lasmezas, PhD, Principal Investigator — Florida Atlantic University
Locations (1):
- FAU Clinical Research Unit, Boca Raton, Florida, United States

IPD SHARING:
Plan to Share IPD: Yes
Primary outcome measure data will be shared.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: IPD and supporting information will be available from June 2027 to Mai 2028.
Access Criteria: The type of analyzes qualifying for data sharing will be those submitted for publication. After publication these data will be freely available. Before publication, a proposal describing planned analyses must be submitted to FAU Office of Research Integrity via the contact information available on the website, and a data sharing agreement must be signed between FAU and the receiving party.